CLINICAL TRIAL: NCT07273760
Title: A Prospective and Observational Study for Effectiveness and Safety Evaluation of VedAryo® (Vedolizumab) in Patients With Inflammatory Bowel Disease
Brief Title: VedAryo® (Vedolizumab) Effectiveness and Safety Evaluation
Status: Completed | Type: Observational
Sponsor: AryoGen Pharmed Co. (Industry)
Responsible Party: Sponsor
Other Study IDs: VDZ.ARY.HV.IV.02
Record Dates: First submitted 2025-11-25; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Ulcerative Colitis (UC); Crohn Disease (CD); Inflammatory Bowel Disease (IBD)
Keywords: vedolizumab; IBD; Ulcerative Colitis; Crohn's disease; Inflammatory Bowel Disease
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Inflammatory Bowel Diseases | interventions — vedolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 52 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants received VedAryo® (Vedolizumab)
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Vedolizumab — Vedolizumab administered IV with a suggested dose of 300 mg at 0, 2, and 6 weeks and then once every 8 weeks

SUMMARY:
The aim of this observational study is to evaluate Effectiveness and safety of VedAryo® (Vedolizumab) in male or female participants with clinical diagnosis of Inflammatory Bowel Disease. The main questions are aim to answer:

1. Is VedAryo® (Vedolizumab) effective in the treatment of Inflammatory Bowel Disease?
2. Is VedAryo® (Vedolizumab) safe in the treatment of Inflammatory Bowel Disease?

In this study, there is no comparison group. Participants received VedAryo® (Vedolizumab)

DETAILED DESCRIPTION:
This research was conducted as a phase IV, post-marketing, observational cohort study, in which VedAryo® (Vedolizumab) was prescribed as part of routine clinical practice, and no study-related intervention was introduced. The study aimed to evaluate the real-world effectiveness and safety of VedAryo® in Iranian patients diagnosed with Inflammatory Bowel Disease (IBD).

The primary objective was to assess the effectiveness of VedAryo® based on clinical response, measured using the Mayo Scoring Index for ulcerative colitis and the Harvey-Bradshaw Index for Crohn's disease during the observation period.

The secondary objective focused on safety, including the incidence of adverse events (AEs) and serious adverse events (SAEs) recorded over the 52-week observational follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Inflammatory bowel disease, including Ulcerative Colitis and Crohn's disease
* Patients with an indication of vedolizumab therapy
* Ability to comprehend and willingness to sign the informed consent form for this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2023-07-16 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-10-05 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Clinical Response at Week 52 | Baseline, week 52
  Clinical response is defined as a decrease from baseline in HBI score of ≥3 points in CD participants and a decrease from baseline in Mayo Score of ≥3 points, ≥30%, and either a decrease from baseline in the rectal bleeding sub score of ≥ 1 or a rectal bleeding sub score of 0 or 1 in UC participants.

SECONDARY OUTCOMES:
Safety Assessment During 52 Weeks | Up to 52 weeks
  Safety assessment, including the incidence of AEs. All AEs are classified based on the Medical Dictionary for Regulatory Activities (MedDRA Desktop Browser 4.0 Beta) terms as System Organ Class (SOC) and Preferred Term (PT). All the reported events are graded according to the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0). Moreover, seriousness of AEs is assessed according to International Council for Harmonisation (ICH-E2B) guidelines. The causality relation is assessed based on the World Health Organization (WHO) criteria.
Percentage of Participants Achieving Clinical Remission at Week 52 | Baseline, week 52
  Clinical remission is defined as a HBI score of <5 points in CD participants and a Mayo Score of ≤2 points and no sub score of >1 in UC participants.

CONTACTS AND LOCATIONS:
Locations (12):
- Iran (12):
  - Dr. Mohammad-Javad Kaviani Clinic, Shiraz, Fars
  - Gilan Gastroenterology and Hepatology Subspecialty Clinic, Rasht, Gilan Province
  - Dr. Ali Beheshti-Namdar Clinic, Mashhad, Razavi Khorasan Province
  - Dr. Hassan Vossoughinia Clinic, Mashhad, Razavi Khorasan Province
  - Dr. Hamid Asadzadeh Aghdaei Clinic, Tehran
  - Dr. Mahtab Shabani Clinic, Tehran
  - Dr. Naser Ebrahimi Daryani Clinic, Tehran
  - Imam Khomeini Hospital, Tehran
  - Mehr Specialty Clinic, Tehran
  - Professor Shahram Agah Gastroenterology, Hepatology, and Endoscopy Subspecialty Clinic, Tehran
  - Shariati Hospital, Tehran
  - Taleghani Hospital, Tehran

IPD SHARING:
Plan to Share IPD: No
Data produced in the present study are available upon reasonable request from the investigators.

REFERENCES:
- [Result] Feagan BG, Rutgeerts P, Sands BE, Hanauer S, Colombel JF, Sandborn WJ, Van Assche G, Axler J, Kim HJ, Danese S, Fox I, Milch C, Sankoh S, Wyant T, Xu J, Parikh A; GEMINI 1 Study Group. Vedolizumab as induction and maintenance therapy for ulcerative colitis. N Engl J Med. 2013 Aug 22;369(8):699-710. doi: 10.1056/NEJMoa1215734. PMID 23964932
- [Result] Yarur A, Mantzaris GJ, Wang S, Adsul S, Kamble P, Cook E, Sajeev G, Guerin A, Bressler B. Stratified Patient Profiling for Vedolizumab Effectiveness in Crohn's Disease: Identifying Optimal Subgroups for Enhanced Treatment Response in the EVOLVE Study. Adv Ther. 2024 Jun;41(6):2324-2341. doi: 10.1007/s12325-024-02825-w. Epub 2024 Apr 24. PMID 38658485
- See also: Related Info — https://link.springer.com/article/10.1007/s12325-024-02825-w